CLINICAL TRIAL: NCT02332538
Title: Randomized Trial Comparing Holmium Laser Enucleation of the Prostate vs. Greenlight 532nm-laser Vapo-Enucleation of the Prostate vs. Bipolar Transurethral Resection of the Prostate in Management of Moderate/Large Benign Prostate Hyperplasia
Brief Title: HoLEP vs. Greenlight 532nm-laser PVEP vs. Bipolar TURP in Management of Moderate/ Large BPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elshal, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS/16.04.79
Record Dates: First submitted 2014-12-27; First posted 2015-01-07 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Benign Prostate Hyperplasia; Lower Urinary Tract Symptoms
Keywords: LASER; PROSTATE; BIPOLAR; HYPERPLASIA; VAPORIZATION
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Greenlight (532nm-laser) PVEP (Active Comparator): 532nm-laser photoselective vapo-enucleation of the prostate)
  Interventions: Procedure: 532nm-laser photoselective vapo-enucleation of the prostate)
- Holmium laser enucleation of prostate (Active Comparator): Holmium-Yag laser enucleation of the prostate
  Interventions: Procedure: Holmium laser enucleation of prostate
- Bipolar TURP (Active Comparator): Bipolar transurethral resection of the prostate in saline
  Interventions: Procedure: Bipolar TURP

INTERVENTIONS:
Procedure: 532nm-laser photoselective vapo-enucleation of the prostate) — using Greenlight (532nm-laser) modified vaporization technique, PVEP (photoselective vapo-enucleation of the prostate)
  Arms: Greenlight (532nm-laser) PVEP
Procedure: Holmium laser enucleation of prostate — Holmium-Yag laser enucleation of the prsotate
  Arms: Holmium laser enucleation of prostate
Procedure: Bipolar TURP — Bipolar transurethral resection of the prostate in saline
  Arms: Bipolar TURP

SUMMARY:
Most guidelines are not strict for recommending single treatment approach for Moderate to large prostate.

In this study the investigators planned to test the Greenlight (532-nm) laser Photoselective Vapo-Enucleation of the Prostate (PVEP) using (XPS) 180W system compared to bipolar transurethral resection of the prostate (TURis) and Holmium Laser Enucleation of the Prostate (HOLEP) in reduction of lower urinary tract symptoms (LUTS) secondary to BPH in a prospective randomized trial.

DETAILED DESCRIPTION:
With a growing body of knowledge on the promising advancements and recent clinical data of the third generations of the Greenlight XPS, it seems to be a real contender in the world of MIS. Contenders of Greenlight laser technology includes bipolar as well as Holmium laser technology.

In this study the investigators planned to test the Greenlight (532-nm) laser Photoselective Vapo-Enucleation of the Prostate (PVEP) using (XPS) 180W system compared to bipolar transurethral resection of the prostate (TURis) and Holmium Laser Enucleation of the Prostate (HOLEP) in reduction of LUTS secondary to BPH in a prospective randomized trial.

Furthermore, all peri-operative parameters, urinary flow parameters, prostate size changes and complications associated with the procedures were compared. The prostate size limitations will be assessed in relation to the outcome measures.

Moderate to large size prostate (80-120 ml TRUS estimated volume) will be randomized to PVEP vs. Bipolar TURP vs. HoLEP.

ELIGIBILITY:
Inclusion Criteria:

1. Patients' age ≥50 years
2. LUTS secondary to BOO due to BPH who failed medical treatment
3. International prostate symptom scores 8 (IPSS) >15 and bother score 8 (QOL) ≥ 3 (according to IPSS question 8)
4. Peak urinary flow rate (Qmax) <15 ml/sec with at least 125 ml voided volume or Patients with acute urine retention secondary to BPH who failed trial of voiding on medical treatment.
5. ASA (American society of anaesthesiologists) score ≤3.
6. TRUS prostate size (>/=80ml)

Exclusion Criteria:

1. Patient with neurological disorder which might affect bladder function as cerebrovascular stroke, Parkinson disease
2. Active urinary tract infection,
3. Presence of active bladder cancer (within the last 2 years)
4. Known prostate cancer patients will be excluded preoperatively on the basis of digital rectal examination, prostate specific antigen level, and TRUS imaging followed by prostate biopsies if necessary.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Re treatment | 3 YEARs
  need for retreatment for recurrent infravesical obstruction following primary surgery

SECONDARY OUTCOMES:
change in symptoms score | 3 year
  degree of improvement in the lower urinary tract symptoms
Urine Flow rate (ml/sec) | 3 year
  degree of improvement in the rate of urine flow

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Elshal, MD, Principal Investigator — Mansoura University
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt